CLINICAL TRIAL: NCT05054205
Title: The Effect on Self-effıcacy of Self-management Program Based on motıvatıonal ıntervıewing in Chronic Obstructive Pulmonary Disease (COPD) patıents: A Randomized Controlled Trial
Brief Title: Motivational Interview-based Self-management Training
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Yeliz Karaçar, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 53043469; HF-18005 (Other Grant/Funding Number: Scientific Research Projects Commission)
Record Dates: First submitted 2021-09-10; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: COPD; Motivational Interviewing; Self Management; Self-Efficacy; Psychiatric Nursing
Keywords: COPD; Motivational interviewing; Self management; Self-Efficacy; Psychiatric nursing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: This randomized controlled experimental study was conducted between March and May 2018 with 39 intervention and 39 control groups, a total of 78 patients in the Chest Diseases Clinic of Chest Diseases Hospital who were treated with COPD. In data collection; ''Patient Data Form'', ''Medical Research Council (MRC) Dyspnea Scale'', ''COPD Self Efficacy Scale (CSES)'' were used.To the experimental group; motivational interview based self-management education was given for 30-45 minutes with groups of 5-8 people, COPD education guide was given, questions were shared with the question-answer method and group interaction was provided. After the self-management education, 3 motivational interviews were conducted 3 days apart with 30-45 minutes. Normal care was continued in the control group. The data were collected in three stages as pre-test, post-test and follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): To the experimental group; motivational interview based self-management education was given for 30-45 minutes with groups of 5-8 people, COPD education guide was given, questions were shared with the question-answer method and group interaction was provided. After the self-management education, 3 motivational interviews were conducted 3 days apart with 30-45 minutes.The data were collected in three stages as pre-test, post-test and follow-up (after 30 day).
  Interventions: Behavioral: Motivational İnterviewing
- Control group (No Intervention): Normal care was continued in the control group.

INTERVENTIONS:
Behavioral: Motivational İnterviewing — The most current version of Motivational İnterviewing (MI) is described in detail in Miller and Rollnick (2013) Motivational Interviewing: Helping people to change (3rd edition). Key qualities include:
  MI is a guiding style of communication, that sits between following (good listening) and directing (giving information and advice).
  MI is designed to empower people to change by drawing out their own meaning, importance and capacity for change.
  MI is based on a respectful and curious way of being with people that facilitates the natural process of change and honors client autonomy.
  Other Names: Self- management training
  Arms: Experimental group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is an important chronic disease that causes increasing mortality and morbidity globally, as well as a social and economic burden. All symptoms (cough, sputum production, etc.), especially dyspnea in COPD, the chronicity of the disease and the need for long-term care limit the lives of the patients. Dyspnea occurring in COPD negatively affects the self-confidence of patients by restricting their activities of daily living, thus causing a decrease in their self-efficacy levels. Low self-efficacy levels cause patients to limit their activities more.

Nurses play an important role in ensuring the management of COPD, supporting patients to continue their activities of daily living, and increasing their self-efficacy levels. Nursing care that includes patient education and counseling is important in providing disease management and symptom control, and increasing the self-efficacy levels of patients. During self-management training, it is necessary to ensure that the patient is an active participant, to use a motivating communication style in the behavior change process and to encourage patients. In this process, it is stated that it is important to use motivational interview techniques in self-management training given by nurses.

DETAILED DESCRIPTION:
This study was conducted to investigate the effect on self-efficacy of self-management education and motivational interview among COPD patients. This randomized controlled experimental study was conducted between March and May 2018 with 39 intervention and 39 control groups, a total of 78 patients in the Chest Diseases Clinic of Chest Diseases Hospital who were treated with COPD. In data collection; ''Patient Data Form'', ''Medical Research Council (MRC) Dyspnea Scale'', ''COPD Self Efficacy Scale (CSES)'' were used. To the experimental group; motivational interview based self-management education was given for 30-45 minutes with groups of 5-8 people, COPD education guide was given, questions were shared with the question-answer method and group interaction was provided. After the self-management education, 3 motivational interviews were conducted 3 days apart with 30-45 minutes. Normal care was continued in the control group. The data were collected in three stages as pre-test, post-test and follow-up. According to the research ethics, self-management education and COPD education guidelines were given to the control group and motivational interviews were conducted. In this study, written consent was obtained from the ethics committee, institutions and patients.

* Self-efficacy levels and dyspnea perception levels of COPD patients are the dependent variables of the study.
* Self-management training and motivational interviewing given to COPD patients are the independent variables of the research.
* Control variables of the study; age, gender, marital status, education status, occupation, employment status, smoking status, duration of being a COPD patient, number of hospitalizations, drug use status, people living with at home, type of warming, participation in COPD education and Pulmonary Rehabilitation program.
* H0: Self-management training and motivational interviewing given to COPD patients have no effect on self-efficacy and dyspnea perception.
* H1: Self-management training and motivational interviewing given to COPD patients have an effect on self-efficacy and dyspnea perception.
* All statistical analyzes were made SPSS 25 package program. The obtained data were analyzed by means of percentage distributions, mean, variance analysis in repeated measures, bonferroni analysis as a further analysis and t test in dependent groups.

ELIGIBILITY:
Inclusion Criteria:

* To receive inpatient treatment with the diagnosis of COPD,
* To be literate,
* To have the cognitive and mental competence to answer questions,
* Disease symptoms are at a level that does not prevent communication

Exclusion Criteria:

* The patient is in an acute exacerbation period,
* Having dyspnea at a level that prevents cooperation,
* Presence of sensory loss related to vision, hearing and speech,
* Presence of cognitive and mental impairment that prevents communication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Self Efficacy | measuring self-efficacy levels at baseline
  COPD Self Efficacy Scale: The scale is composed of 34 items. It is a five-point Likert scale; one corresponds to 'I am not confident' (not efficacious), two 'I am a little confident' (efficacious), three 'I am confident to some extent' (efficacious), four 'I am quite confident' (efficacious) and 5 'I am very confident' (efficacious). The highest and lowest scores for the scale are 170 and 34, respectively. An increase in the self-efficacy scale mean score indicates that the patient's self-efficacy level has improved. Total or mean scores for the scale and its subscales are utilized for the evaluation of self-efficacy in patients with COPD.
Self Efficacy | Change in self-efficacy level immediately after completion of a two-week motivational interview-based self-management training
  COPD Self Efficacy Scale: The scale is composed of 34 items. It is a five-point Likert scale; one corresponds to 'I am not confident' (not efficacious), two 'I am a little confident' (efficacious), three 'I am confident to some extent' (efficacious), four 'I am quite confident' (efficacious) and 5 'I am very confident' (efficacious). The highest and lowest scores for the scale are 170 and 34, respectively. An increase in the self-efficacy scale mean score indicates that the patient's self-efficacy level has improved. Total or mean scores for the scale and its subscales are utilized for the evaluation of self-efficacy in patients with COPD.
Self Efficacy | Change in self-efficacy level one month after motivational interview-based self-management training
  COPD Self Efficacy Scale: The scale is composed of 34 items. It is a five-point Likert scale; one corresponds to 'I am not confident' (not efficacious), two 'I am a little confident' (efficacious), three 'I am confident to some extent' (efficacious), four 'I am quite confident' (efficacious) and 5 'I am very confident' (efficacious). The highest and lowest scores for the scale are 170 and 34, respectively. An increase in the self-efficacy scale mean score indicates that the patient's self-efficacy level has improved. Total or mean scores for the scale and its subscales are utilized for the evaluation of self-efficacy in patients with COPD.

SECONDARY OUTCOMES:
Perception of dyspnea | Measuring perception of dyspnea levels at baseline
  Medical Research Council Dyspnea Scale: The Medical Research Council Dyspnea Scale is a 0-4 point category scale in which one of five expressions related to the perception of dyspnea is selected to best describe the patient's dyspnea level. ''0 points'' no dyspnea ''4 points'' indicates very severe dyspnea.
Perception of dyspnea | Change in perception of dyspnea level immediately after completion of a two-week motivational interview-based self-management program
  Medical Research Council Dyspnea Scale: The Medical Research Council Dyspnea Scale is a 0-4 point category scale in which one of five expressions related to the perception of dyspnea is selected to best describe the patient's dyspnea level. ''0 points'' no dyspnea ''4 points'' indicates very severe dyspnea.
Perception of dyspnea | Change in perception of dyspnea level one month after motivational interview-based self-management training
  Medical Research Council Dyspnea Scale: The Medical Research Council Dyspnea Scale is a 0-4 point category scale in which one of five expressions related to the perception of dyspnea is selected to best describe the patient's dyspnea level. ''0 points'' no dyspnea ''4 points'' indicates very severe dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Karaçar, M.Sc., Principal Investigator — Denizli Buldan Chest Diseases Hospital
Locations (1):
- Denizli Buldan Chest Diseases Hospital, Denizli, Buldan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2018. Available from: http://goldcopd.org.
- [Background] Miller WR, Rollnick S. Motvational Interviewing. Motivasyonel Görüşme İnsanları Değişime Hazırlama. Karadağ F, Ögel K, Tezcan AE. (Ed), HYB Basım Yayın Matbaası, Ankara, 2009, 216-231.
- [Result] Benzo R, Vickers K, Ernst D, Tucker S, McEvoy C, Lorig K. Development and feasibility of a self-management intervention for chronic obstructive pulmonary disease delivered with motivational interviewing strategies. J Cardiopulm Rehabil Prev. 2013 Mar-Apr;33(2):113-23. doi: 10.1097/HCR.0b013e318284ec67. PMID 23434613
- [Result] Abedi HA, Salimi S, Feizi A, et al. Assessment of relationship between self-efficacy and self-care in COPD Patients. Journal of Urmia Nursing and Midwifery Faculty, 2012, 10(1), 68-74.
- [Result] Celli BR, Decramer M, Wedzicha JA, Wilson KC, Agusti A, Criner GJ, MacNee W, Make BJ, Rennard SI, Stockley RA, Vogelmeier C, Anzueto A, Au DH, Barnes PJ, Burgel PR, Calverley PM, Casanova C, Clini EM, Cooper CB, Coxson HO, Dusser DJ, Fabbri LM, Fahy B, Ferguson GT, Fisher A, Fletcher MJ, Hayot M, Hurst JR, Jones PW, Mahler DA, Maltais F, Mannino DM, Martinez FJ, Miravitlles M, Meek PM, Papi A, Rabe KF, Roche N, Sciurba FC, Sethi S, Siafakas N, Sin DD, Soriano JB, Stoller JK, Tashkin DP, Troosters T, Verleden GM, Verschakelen J, Vestbo J, Walsh JW, Washko GR, Wise RA, Wouters EF, ZuWallack RL; ATS/ERS Task Force for COPD Research. An Official American Thoracic Society/European Respiratory Society Statement: Research questions in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2015 Apr 1;191(7):e4-e27. doi: 10.1164/rccm.201501-0044ST. PMID 25830527
- [Result] Chen SM, Creedy D, Lin HS, Wollin J. Effects of motivational interviewing intervention on self-management, psychological and glycemic outcomes in type 2 diabetes: a randomized controlled trial. Int J Nurs Stud. 2012 Jun;49(6):637-44. doi: 10.1016/j.ijnurstu.2011.11.011. Epub 2011 Dec 30. PMID 22209215
- [Result] Emme C, Mortensen EL, Rydahl-Hansen S, Ostergaard B, Phanareth K. Danish version of 'The COPD self-efficacy scale': translation and psychometric properties. Scand J Caring Sci. 2012 Sep;26(3):615-23. doi: 10.1111/j.1471-6712.2011.00963.x. Epub 2012 Jan 24. PMID 22272564
- [Result] World Health Organization. (2018). The top 10 causes of death. https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death (26 Mayıs 2018).